CLINICAL TRIAL: NCT02482376
Title: A Phase II Preoperative Single-Fraction Partial Breast Radiotherapy in Early Stage Breast Cancer: Analysis of Pathologic Response
Brief Title: Preoperative Single-Fraction Radiotherapy in Early Stage Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00063848
Record Dates: First submitted 2015-06-22; First posted 2015-06-26 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm 21Gy stereotactic radiotherapy (Other): Subjects will receive a single fraction of 21Gy of stereotactic radiotherapy before proceeding to surgery.
  Interventions: Radiation: Stereotactic body radiotherapy ( SBRT)

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy ( SBRT) — Single fraction of 21 Gy stereotactic radiotherapy (SBRT)delivered pre-operatively to subjects with early stage breast cancer
  Other Names: SBRT

SUMMARY:
This protocol seeks to build on the favorable results of the investigators' phase I trial (Pro00015617) by extending the findings to a larger cohort of subjects.In this study, the investigators hypothesize that 21Gy (Gray) as a single fraction can be delivered preoperatively to a larger group of subjects (n100).

The primary objective is to determine physician reported rates of good/excellent cosmesis at baseline and 6 months, 1, 2, and 3 years post-treatment as measured by the NRG cosmesis scale

DETAILED DESCRIPTION:
The study team hypothesizes that a single fraction of 21Gy can be delivered preoperatively to the intact breast tumor with acceptable cosmetic outcomes. Furthermore, the investigators anticipate that pre- and post-radiation breast tumor samples will provide an avenue for understanding breast cancer radiation response

Rationale for single-fraction preoperative technique

This trial is proposed to build on the favorable results of the investigators' phase I trial by extending the findings to a larger cohort of subjects. The preoperative approach has several advantages:

1. a small intact breast tumor results in significantly less uninvolved breast tissue receiving high radiation doses which likely decreases toxicity;
2. more accurate targeting of the high-risk areas of subclinical disease surrounding the tumor is possible,
3. smaller treatment volumes are amenable to dose escalation which can further accelerate treatment and improve accessibility for subjects,
4. this technical approach is widely utilized in other tumor sites and can be delivered at most radiation facilities
5. the pre-operative approach provides a novel opportunity to study breast cancer radiation response.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a biopsy proven diagnosis of ductal carcinoma in situ or invasive carcinoma of the breast

   a. Biopsy tissue (either slides or block) from outside institutions will be reviewed to confirm diagnosis.
2. Breast preservation candidates (no prior breast or nodal radiotherapy, no imaging evidence of multicentric or multifocal disease, no pregnant women, and no comorbid conditions precluding surgery)
3. Clinical T1N0M0 invasive carcinoma or Ductal carcinoma in situ (DCIS) < or equal to 2cm
4. 60 years of age or older or 50-59 with a low Oncotype score (0-17) Oncotype is not required for women diagnosed with DCIS.
5. Estrogen receptor positive (ER+), Human epidermal growth factor 2 negative (HER2-) HER-2 status is not required for women diagnosed with DCIS.
6. Women of child-bearing potential must consent to use adequate contraception during the course of the study. Female subjects must agree to use a medically acceptable contraceptives including: (1) surgical sterilization (such as a tubal ligation or hysterectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD). Contraceptive measures such as Plan B (TM), sold for emergency use after unprotected sex, are not acceptable methods for routine use.
7. White blood cells (WBC) > 3000, Hemoglobin ( Hgb) > 9, platelets >100000 within 30 days of consent
8. Eligible for contrasted magnetic resonance imaging (MRI) on initial evaluation with glomerular filtration rate (GFR) ≥ 60 ml/min. A diagnostic MRI ordered within one month will be considered an acceptable alternative and will not be repeated.
9. Outside breast imaging will be reviewed at Duke to confirm findings are consistent with trial eligibility.

Exclusion Criteria:

1. Neoadjuvant chemotherapy
2. Breast implant in the breast to be treated with SBRT
3. Medical conditions that may increase risk for poor cosmetic outcome (i.e. Lupus, rheumatoid arthritis, scleroderma)
4. Subjects unable to receive study treatment planning secondary to body habitus or inability to lie flat on the stomach at length
5. HER2 positive
6. Positive serum pregnancy test
7. Insufficient breast imaging to judge clinical stage
8. Subjects without placement of a biopsy clip at the diagnostic procedure who are unwilling to undergo clip placement.
9. Subjects in whom treatment planning constraints cannot be met

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2032-03-10 (Estimated)

PRIMARY OUTCOMES:
Physician reported rates of good/excellent cosmesis. | Through study completion estimated to be 3 years
  Physician will independently complete the physician NRG Oncology cosmesis scale at the designated time points

SECONDARY OUTCOMES:
Ki-67 will be assessed as a measure of tumor response | Through study completion estimated to be 3 years
  Ki-67 will be assessed in the pre and post radiotherapy tissue samples
Patient reported rates of good/excellent cosmesis | Through study completion estimated to be 3 years
  Patients will independently complete the patient NRG Oncology cosmesis scale at designated timepoints
The impact of radiation on gene expression | Through study completion estimated to be 3 years
  Gene expression will be assessed using the Affymetrix Human Transcriptome Array (HTA) arrays designed for formalin fixed paraffin embedded (FFPE) samples on pre and post radiation therapy tissue samples.
Local control in the treated breast relative to historic controls | Through study completion estimated to be 5-10 years
  Annual clinical examination combined with breast imaging
Assess the impact of RT on circulating cell free DNA | Through study completion estimated to be 3 years
  Oxidative stress biomarkers will be measured in serum and urine collected at the same timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Blitzblau, MD PhD, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States